CLINICAL TRIAL: NCT01361867
Title: Robotic Assessment of Lower Extremity Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-P-002030
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy Subjects
Keywords: motor adaptation; lower extremity motor learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robot-induced perturbations (Other): The subject walks on a treadmill with his/her legs strapped to a robotic system (Lokomat by Hocoma AG) that generates mechanical perturbations aimed to modify the subject's walking pattern.
  Interventions: Device: Robot-induced perturbations

INTERVENTIONS:
Device: Robot-induced perturbations — A robotic system is used to generate mechanical perturbations and study how subjects generate motor adaptations in response to the mechanical perturbations.

SUMMARY:
The aim of the study is to assess the ability of healthy subjects to generate a motor adaptation in response to a mechanical perturbation generated by a robotic system for treadmill-based gait training (Lokomat by Hocoma AG, a device that received 510K FDA clearance).

DETAILED DESCRIPTION:
The study is divided into two phases.

In phase I of the study, we intend to assess the response of individuals to a variety of different mechanical perturbations generated by a robotic system for treadmill-based gait training (Lokomat by Hocoma AG). Such response is quantified as a displacement from the baseline (i.e. gait cycles with no mechanical perturbation) trajectory of motion of the foot during the swing phase of the gait cycle. This portion of the study is expected to allow us to identify mechanical perturbations that are suitable to study motor adaptation.

In phase II of the study, we plan to carry out experiments using the above-mentioned robotic system to assess the magnitude of the motor adaptation to the mechanical perturbations identified in phase I as suitable for the study. The magnitude of the motor adaptation is quantified as the percentage of the deviation from the baseline trajectory of motion of the foot that subjects compensate for when exposed to the perturbation during multiple consecutive gait cycles.

It is worth noticing that the robotic system utilized to generate the mechanical perturbations (i.e. Lokomat by Hocoma AG) is not programmed by the company to generate the mechanical perturbations evaluated in this project. Our research group wrote the programs to generate such perturbations. It is also worth emphasizing that the 510K FDA clearance does not cover the modifications implemented by our research group.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, healthy adults age 18-55 years, with normal gait.

Exclusion Criteria:

* Lower extremity fractures
* Current or previous history of orthopedic injury that would prevent safe use of the robotic system
* Body/femoral length size beyond the limits of robotic system (femur length between 350-470mm)
* Body weight > 135kg (~298 lbs) maximum limit of the body weight support system
* Skin lesions on the lower extremities
* Cardiovascular or pulmonary contraindications
* Motor system or proprioceptive impairments
* Severe cognitive impairments that would prevent the use of the robotic system

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited by posting flyers in public areas and by contacting subjects who had previously expressed interest for volunteering in research studies in our laboratory.
Period: Overall Study
Arm/Group | Robot-induced Perturbations
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot-induced Perturbations
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Step Length [Mean (Standard Deviation); unit: cm] — Please notice that step length was defined as the maximum value of the foot position in the anteroposterior direction in a coordinate system positioned at the center of rotation of the robotic joint connecting the pelvis and thigh components of the exoskeleton system. In other words, this measure differs from standard measures of step length during overground walking.
  cm | 25.0 (0.3)
Step Height [Mean (Standard Deviation); unit: cm] — Please notice that step height was defined as the distance between the foot and the belt of the treadmill during the midswing phase of the gait cycle. This definition of step height allowed us to measure it where the effect of the perturbation led to a maximum deviation from the baseline value
  cm | 9.7 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Step Length Adaptation
Description: The percentage of the step length change caused by the mechanical perturbation that subjects compensate for
Time Frame: within a trial of the experiment (i.e. a few minutes)
Measure: Mean (Standard Error); unit: % of step length compensated for
Arm/Group | Robot-induced Perturbations
Number analyzed (Participants) | 15
% of step length compensated for | 83.6 (4.5)

2. Secondary Outcome: Step Height Adaptation
Description: The percentage of the step height change caused by the mechanical perturbation that subjects compensate for
Time Frame: within a trial of the experiment (i.e. a few minutes)
Measure: Mean (Standard Error); unit: % step height compensated for
Arm/Group | Robot-induced Perturbations
Number analyzed (Participants) | 15
% step height compensated for | 6.1 (4.1)

ADVERSE EVENTS:
Time Frame: Through study completion (three sessions over a period of one week).
Arm/Group | Robot-induced Perturbations
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The study was based on pilot experiments (N=35) aimed to determine how to use the robot to perturb step length and step height during gait. In the actual study (N=15), the investigators assessed how individuals adapted to the perturbations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No